CLINICAL TRIAL: NCT05157633
Title: Oral Exploration of Objects and Food Diversification
Acronym: OPENING
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: OPENING
Record Dates: First submitted 2021-09-08; First posted 2021-12-15 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Infant Development
Keywords: Infants and children with eating difficulties

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Children without eating difficulties
  Interventions: Other: Controls
- Patients: Children with eating difficulties

INTERVENTIONS:
Other: Controls — questionnaire food scale: HME data collection of food survey
  Groups: Controls

SUMMARY:
Eating difficulties in infants and young children are defined as all the difficulties in feeding oneself in an appropriate and satisfactory manner. These disorders affect approximately 20 to 25% of infants and young children, and thus constitute one of the most frequent reasons for consultation in these age groups. Many of these children continue to be received in consultation.

Studies show that the lack of intraoral exploration in children could be associated with later difficulties in accepting different textures or new foods. Our clinical examination of sensorimotor functions shows signs of sensory hyper reactivity that are very common in children who always wipe their hands when in contact with food or sticky objects and for those who experience difficulty in brushing or grooming themselves.

In all of the publications available which includes pubmed, there is no mention of the lack of exploration of objects and the stigma of sensory hyper-responsiveness even if this latter was not entirely detailed in the descriptions made.

The trial hypothesis is that this exploration defect corresponds to early sensory hyperreactivity which also plays a deleterious role in the acceptance of new textures and new foods.

In this trial we propose a comparison study with a controlled population of children without eating difficulties as defined by the Montreal MCH score to validate a statistical link between the difficulties in food diversification beyond 18 months and the lack of exploration of the environment with 'mouthing' between 6 and 10 months.

Investigators will analyse consultation questionnaires dedicated to eating difficulties retrospectively (patients) and will compare them with questionnaires of children from daycares without eating difficulties (controls).

DETAILED DESCRIPTION:
To conduct this study the controls will be recruited from daycares and different nursery schools after agreement with the heads of establishments.

Two questionnaires along with an information note will be distributed to the parents and will be completed in a non-identifying manner, retrieved by the teachers and then sent to the principal investigator.

The questionnaires include the validated Montreal HME questionnaire which will detect the possible existence of eating difficulties and a more general questionnaire on the psychomotor development of the child (not validated because a qualitative questionnaire without a score). The collection of data will be prospective for controls.

Patients on the other hand will be recruited retrospectively from the dedicated oral consultation at the Hospital.

ELIGIBILITY:
Inclusion Criteria:

* For patients: Children aged between 9 months and 6 years with eating difficulties defined by the Montreal HME score> = 61.

For controls: children aged between 9 months and 6 years attending a crèche who agreed to participate in the study.

Not opposing participation in the study.

Exclusion Criteria:

Exclusion of controls who have:

* an eating disorder defined by an MCH score> = 61 (score defined for the inclusion criteria)
* encephalopathy, neuro-metabolic disorder, genetic syndrome (after response to the questionnaire)

For patients and controls:

* Encephalopathies
* Neuro-metabolic disorders
* Suspected or identified genetic syndromes

Ages: 9 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with eating difficulties and children from nurseries without eating difficulties (controls).
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with a delay or lack of acquisition of oral exploration of objects. | 1 day
  Deferred presence or absence of the acquisition of the competence of oral exploration of objects between 6 and 10 months by a qualitative questionnaire without score not validated

SECONDARY OUTCOMES:
To determine if there is a link between the inability to orally explore objects and difficulties in seeing and/or touching and/or smelling certain types of food | 1 day
  Number of children with difficulty seeing and / or touching and / or smelling certain types of food and an inability to explore objects orally.
To determine if there is a link between the inability to orally explore objects and difficulties in seeing and/or touching and/or smelling certain types of food | 1 day
  Percentage of children with difficulty seeing and / or touching and / or smelling certain types of food and an inability to explore objects orally.
To determine if there is a link between the inability to orally explore objects and the inability to touch certain non-food textures | 1 day
  Number of children with an inability to touch certain non-food textures and an inability to orally explore objects by a qualitative questionnaire without score not validated
To determine if there is a link between a link between the inability to orally explore objects. And the inability to touch certain non-food textures | 1 day
  percentage of children with an inability to touch certain non-food textures and an inability to orally explore objects
To determine if there is a link between a link between the inability to orally explore objects and the absence of crawling in motor development. | 1 day
  Number and percentage of children who have crawled in their psychomotor development
To determine if there is a link between a link between the inability to orally explore objects and the absence of crawling in motor development. | 1 day
  Number of children who orally explored the objects
To determine if there is a link between a link between the inability to orally explore objects and the absence of crawling in motor development. | 1 day
  percentage of children who orally explored the objects
To determine if there is a link between an incidence of constipation in both groups of children | 1 day
  Number of children with constipation according to ROME IV criteria
To determine if there is a link between an incidence of constipation in both groups of children | 1 day
  percentage of children with constipation according to ROME IV criteria

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Robert Debré, 48 Bd Sérurier, Paris, France

IPD SHARING:
Plan to Share IPD: No